CLINICAL TRIAL: NCT00362505
Title: An Open-label, Phase III Clinical Trial to Evaluate the Safety and Antiviral Activity of Clevudine in Chronic Hepatitis B Patients Who Have Completed the L-FMAU-301 or L-FMAU-302 Trials
Brief Title: Safety and Antiviral Activity of Clevudine in Patients Who Have Completed the L-FMAU-301 or L-FMAU-302 Trials
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L-FMAU-303
Record Dates: First submitted 2006-08-08; First posted 2006-08-10 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2006-06

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — clevudine

INTERVENTIONS:
Drug: Clevudine

SUMMARY:
The purpose of this study is to determine safety and efficacy of clevudine 10 mg qd for 24 weeks after completion of 24-week treatment with clevudine 30 mg qd with 12 weeks follow-up period

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between 18 and 60, inclusive
2. Patients who have completed L-FMAU-301 or L-FMAU-302 clinical trial.
3. Patient is HBsAg positive at week 48 in L-FMAU-301 or L-FMAU-302.
4. Patient has bilirubin levels less than 2.0 mg/dL, prothrombin time of less than 1.7 (INR), a serum albumin level of at least 3.5 g/dL at week 48 in L-FMAU-301 or L-FMAU-302.
5. Women of childbearing potential must have a negative serum (β-HCG) pregnancy test at screening.
6. Patient is able to give written informed consent prior to study start and to comply with the study requirements.

Exclusion Criteria:

1. Patients with HBV DNA < 4,700 copies/mL, ALT normalization and consecutive e seroconversion at week 40 and 48 in L-FMAU-301
2. Patients with HBV DNA < 4,700 copies/mL and ALT normalization in L-FMAU-302
3. Patient is currently receiving antiviral, immunomodulatory or corticosteroid therapy.
4. Patients previously treated with α-interferon, lamivudine, lobucavir, adefovir or any other investigational nucleoside for HBV infection.
5. Patient has a history of ascites, variceal hemorrhage or hepatic encephalopathy.
6. Patient is coinfected with HCV, HDV or HIV.
7. Patient with clinical evidence of liver mass or hepatocellular carcinoma and α-Fetoprotein > 50 ng/mL
8. Patient is pregnant or breast-feeding.
9. Patient is unwilling to use an "effective" method of contraception during the study and for up to 3 months after the use of study drug ceases. For males, condoms should be used. Females must be surgically sterile (via hysterectomy or bilateral tubal ligation) or post-menopausal or using at least medically acceptable barrier method of contraception (i.e. IUD, barrier methods with spermicide or abstinence)
10. Patient has a clinically relevant history of abuse of alcohol or drugs.
11. Patient has a significant gastrointestinal, renal, hepatic (decompensated), bronchopulmonary, biliary diseases excluding asymptomic GB stone, neurological, cardiovascular, oncologic or allergic disease. The patient with a benign tumor except for liver mass, excluded if judged by an investigator that the continuation of study would be interfered by the tumor.
12. Patient has creatinine clearance less than 60mL/min as estimated by the following formula:

(140-age in years) (body weight [kg])/(72)(serum creatinine [mg/dL]) [Note: multiply estimates by 0.85 for women]

13.Patient whom investigator consider is not suitable in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-06; Study Completion 2006-03

PRIMARY OUTCOMES:
Efficacy:change from baseline in HBV DNA; Safety: clinically measured adverse events, abnormality of laboratory tests and abnormality of vital signs, ECG.

SECONDARY OUTCOMES:
Efficacy:; Proportion of patients with HBV DNA below the assay Limit of Detection; Proportion of patients with HBeAg loss and/or seroconversion (HBeAg loss and HBeAb gain); Proportion of ALT normalization

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Suk Lee, MD. PhD, Principal Investigator — Seoul National University Hospital
Locations (32):
- South Korea (32):
  - Pusan National University Hospital, Ami-dong, Seo-gu, Busan
  - Kosin Medical Center, Amnam-dong, Seo-gu, Busan
  - Pusan Paik Hospital, Gaegeum-dong, Busan
  - Chungnam National University Hospital, Daesa-dong, Jung-gu, Daechon
  - Yeungnam University Medical Center, Daemyoung-dong, Nam-gu, Daegu
  - Keimyumg University Dongsan Medical Center, Jung-gu,, Daegu
  - Kyungpook National University Medical Hospital, Jung-gu, Daegu
  - Korea University Guro Hospital, Seoul, Guro-gu
  - Chonnam National University Hospital, Hak-1-dong, Dong-gu, Gwangju
  - St. Mercy's Hospital, Bupyoung-dong, Bupyoung-gu, Incheon
  - Inha University Hospital, Sinhung-dong, Jung-gu, Incheon
  - Wonkwang University Hospital, Iksan, Jeollabuk-do
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Seoul National University Hospital, Seoul, Jongno-Gu
  - National Cancer Center, Ilsan-gu, Kyounggi-do
  - St. Holly Family Mary's Hospital, Puch’un, Kyounggi-do
  - Pochon CHA University Hospital, Seongnam-gu, Kyounggi-do
  - Gil Medical Center, Incheon, Namdong-Gu
  - Korea University Anam Hospital, Anam-dong, Sungbuk-ku, Seoul
  - KangNam St. Mary's Hospital, Banpo-dong, Seocho-gu, Seoul
  - Kangnam Sacred Heart Hospital, Daelim-dong, Yongdeungpo-gu, Seoul
  - Yongdong Severance Hospital, Dogok-dong, Kangnam-gu, Seoul
  - Korea Cancer Center Hospital, Gongneung-dong, Nowon-gu, Seoul
  - Soon Chun Hyang University Hospital, Hannam-dong, Yongsan-gu, Seoul
  - Samsung Medical Center, Ilwon-dong, Songpa-gu, Seoul
  - Seoul Paik Hospital, Jeo-dong, Seoul
  - Ehwa Womans University Mokdong Hospital, Mok-dong, Yangcheon-gu, Seoul
  - Seoul Asan Medical Center, Pungnap-dong, Kangnam-gu, Seoul
  - Kangbuk Samsung Hospital, Pyoung-dong, Chongro-gu,, Seoul
  - Severance Hospital, Shinchon- Dong, Seodaemun-gu, Seoul
  - St. Vincent's Hospital, Ji-dong,, Paldal-gu, Suwon
  - St. Mary's Hospital, Seoul, Yungdungpo-Gu